CLINICAL TRIAL: NCT02250924
Title: Caffeinated Gum to Prevent Post-Operative Ileus: A Prospective, Randomized, Placebo-controlled Trial
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Investigator decision - clinical practice change
Sponsor: The Guthrie Clinic (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Supportive Care
Other Study IDs: GC1410-55
Record Dates: First submitted 2014-09-22; First posted 2014-09-26 (Estimated); Last update posted 2020-06-04 (Actual); Status verified 2020-06

CONDITIONS: C.Surgical Procedure; Digestive System
MeSH Terms: interventions — Caffeine; Chewing Gum

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Placebo (Placebo Comparator): Subjects will wear a silicone bracelet for 30 minutes 3 times daily at 8 am, 12 pm and 4 pm.
  Interventions: Behavioral: wear silicone bracelet
- Sugar-less Gum (Sham Comparator): Subjects will chew one stick of sugar-less gum for 30 minutes 3 times daily at 8 am, 12 pm and 4 pm.
  Interventions: Other: Gum
- Caffeinated Gum (Experimental): Subjects will chew one stick of caffeinated gum (100mg caffeine per stick) for 30 minutes 3 times daily at 8 am, 12 pm and 4 pm.
  Interventions: Dietary Supplement: Caffeine; Other: Gum

INTERVENTIONS:
Dietary Supplement: Caffeine — caffeinated gum
  Arms: Caffeinated Gum
Other: Gum — Chewing gum
  Arms: Caffeinated Gum; Sugar-less Gum
Behavioral: wear silicone bracelet — Subjects will put on bracelet to correspond with times for chewing gum
  Arms: Placebo

SUMMARY:
This is a randomized, three-arm, double-blind, placebo-controlled, Phase III clinical trial of caffeinated gum and sugar-less gum in adult patients after an abdominal procedure. Patients will be randomized to receive placebo, sugar-less gum or caffeinated gum three times daily for 30 minutes starting the day following surgery until discharge or 24 hours after attainment of the primary endpoint.

ELIGIBILITY:
Inclusion Criteria:

* Abdominal procedure (Laparoscopic or open, occurring electively), American Society of Anesthesiologists (ASA) physical status score ≤ 3, Glasgow Coma Score (GCS) ≥ 15.

Exclusion Criteria:

* ASA physical status score of >3, GCS < 15, complete bowel obstruction, history of cardiac arrhythmia, history of phenylketonuria, alcohol abuse. substance abuse dentures

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2017-01 (Estimated); Primary Completion 2020-05 (Actual); Study Completion 2020-05-28 (Actual)

PRIMARY OUTCOMES:
Mean time to GI function recovery (GI-3) | An expected average of 5 days

SECONDARY OUTCOMES:
Mean length of postoperative hospitalization | Up to 30 days
Rate of postoperative ileus | Up to 30 days
Adverse event rates | Up to 30 days postoperative

CONTACTS AND LOCATIONS:
Overall Officials: Karim Sadik, MD, Principal Investigator — The Guthrie Clinic
Locations (1):
- The Guthrie Clinic, Sayre, Pennsylvania, United States